CLINICAL TRIAL: NCT01920477
Title: OPV116910: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Investigate the Efficacy and Safety of Ofatumumab Injection for Subcutaneous Use in Subjects With Pemphigus Vulgaris
Brief Title: Efficacy and Safety of Ofatumumab in Treatment of Pemphigus Vulgaris
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Novartis has acquired the rights to ofatumumab and terminated the OPV116910 and OPV117059 studies. This decision is not linked to any safety consideration.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116910
Record Dates: First submitted 2013-07-03; First posted 2013-08-12 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-05

CONDITIONS: Pemphigus Vulgaris
Keywords: Pemphigus; MAB; autoimmune disorder; human CD20 antigen; subcutaneous; vulgaris; Phase 3; monoclonal antibody; ofatumumab; PV; rare disease; OMB157; adult
MeSH Terms: conditions — Pemphigus; Autoimmune Diseases; Rare Diseases | interventions — ofatumumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ofatumumab (Experimental): Subject received subcutaneous administration of ofatumumab 20 mg once every 4 weeks through Week 56, with an additional 20 mg dose (that is 40mg total) at both Week 0 and Week 4.
  Interventions: Biological: Ofatumumab
- Placebo (Placebo Comparator): Subject received subcutaneous administration of matching placebo of ofatumumab once every 4 weeks through Week 56, with an additional dose at both Week 0 and Week 4.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ofatumumab — Ofatumumab (human monoclonal antibody) was provided in prefilled glass syringes initial syringes contained 0.6ml (60mg) of concentration 100 mg/m: drug product subsequently modified to 0.4 mL (20mg) concentration (50mg/ML) drug product
  Arms: Ofatumumab
Biological: Placebo — Placebo to match the active doses will consist of prefilled glass syringes filled with normal saline.
  Arms: Placebo

SUMMARY:
Pemphigus vulgaris (PV) is a rare, chronic, debilitating, and potentially life-threatening autoimmune disorder that is characterized by mucocutaneous blisters. Ofatumumab is a novel monoclonal antibody (mAb) that specifically binds to the human CD20 antigen, which is expressed only in B lymphocytes.

The purpose of this study was to evaluate the efficacy, tolerability, and safety of ofatumumab injection for subcutaneous use (ofatumumab SC) 20 milligrams (mg) administered once in every 4 weeks, (with an additional 20 mg loading dose [i.e. 40 mg total] at both Week 0 and Week 4) in subjects with PV. It was anticipated that with sustained B-cell depletion in the presence of ofatumumab SC, and the resultant reduction of pathogenic anti Dsg (desmoglein) autoantibodies in PV, that clinical remission of the disease would result.

DETAILED DESCRIPTION:
Novartis terminated the development of the PV program and this study was terminated for non-safety reasons

ELIGIBILITY:
Inclusion criteria

* Adults (18 through 70 years of age) with clinically-documented diagnosis of PV for >2 months and <10 years.
* History of biopsy consistent with PV (Hematoxylin and Eosin staining and direct immunofluorescence). If no history, a biopsy may be performed during the Screening Period.
* At least 1 previous episode of a failed steroid taper (ie, disease flare/relapse) at a prednisone/prednisolone dose >10 mg/day. The following criteria must have been met as evidence of disease severity at the time of the failed steroid taper: a) A Pemphigus Severity of Clinical Disease score of moderate (2) or severe (3) (may be historical/retrospective assessment). b) Required a treatment change at the time of the failed steroid taper of at least one of the following: i) A steroid increase to >=20 mg/day OR ii) The addition of immunosuppressive/immunomodulatory agent/treatment OR iii) A dose increase of immunosuppressive/immunomodulatory agent/treatment
* Screening anti-Dsg antibodies consistent with a diagnosis of PV (ie, elevated antiDsg3 antibodies).
* Has initiated and received a stable dose of prednisone/prednisolone from a minimum of 20 mg/day (example: 0.25 mg/kg/day for an 80 kg person) up to a maximum of 120 mg/day or 1.5 mg/kg/day (whichever is higher) for >=2 weeks prior to randomization.
* Has exhibited PV disease control, defined as no new lesions for >=2 weeks.
* A female subject is eligible to enter the study if she: Is of non-child bearing potential, who is either surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or post-hysterectomy) or is postmenopausal without menses for >2 years. Women who are <2 years postmenopausal are required to have menopausal status confirmed by follicle-stimulating hormone (FSH) and estradiol levels at the screening evaluation. If FSH and estradiol levels do not provide confirmation of menopause, subject will be considered to be of childbearing potential.

Exclusion Criteria:

* Diagnosis of pemphigus foliaceus, paraneoplastic pemphigus, or other autoimmune blistering disease (other than pemphigus vulgaris).
* Past or current history of hypersensitivity to components of the investigational product or medically significant adverse effects (including allergic reactions) from cetirizine (or antihistamine equivalent) or paracetamol/acetaminophen.
* Prior treatment with rituximab without achieving disease control within 6 months of initiating rituximab dosing.
* Prior treatment with immunosuppressant or immunomodulation agents within the protocol specified periods
* Evidence or history of clinically significant infections

For Japan: Evidence or history of clinically significant infection or medical condition including: Pneumocystis pneumonia or interstitial pneumonia

* Past or current malignancy, except for cervical carcinoma Stage 1B or less, noninvasive basal cell and squamous cell skin carcinoma and cancer diagnoses with a duration of complete response (remission) >5 years
* Significant concurrent, uncontrolled medical condition that could affect the subject's safety, impair the subject's reliable participation in the study, impair the evaluation of endpoints, or necessitate the use of medication not allowed by the protocol. This includes subjects who require any systemic steroid treatment for a concurrent medical condition (other than pemphigus vulgaris).
* Use of an investigational drug or other experimental therapy within 4 weeks, 5 pharmacokinetic half-lives, or the duration of biological effect (whichever is longer) prior to Screening.
* Electrocardiogram (ECG) showing a clinically significant abnormality or showing a QTc interval ≥450 msec (≥480 msec for subjects with a bundle branch block)
* Woman who is breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (7):
  - Novartis Investigational Site, Los Angeles, California
  - Novartis Investigational Site, Atlanta, Georgia
  - Novartis Investigational Site, Ann Arbor, Michigan
  - Novartis Investigational Site, Buffalo, New York
  - Novartis Investigational Site, Durham, North Carolina
  - Novartis Investigational Site, Pittsburgh, Pennsylvania
  - Novartis Investigational Site, Salt Lake City, Utah
- Australia (2):
  - Novartis Investigational Site, East Melbourne, Victoria
  - Novartis Investigational Site, Melbourne, Victoria
- Novartis Investigational Site, Thessaloniki, Greece
- Israel (2):
  - Novartis Investigational Site, Ramat Gan
  - Novartis Investigational Site, Tel Aviv
- Novartis Investigational Site, Milan, Lombardy, Italy
- Novartis Investigational Site, Tokyo, Japan
- Novartis Investigational Site, Warsaw, Poland
- Novartis Investigational Site, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-nine subjects were screened.
Groups:
- Ofatumumab: Subject will receive subcutaneous administration of ofatumumab 20 mg once every 4 weeks through Week 56, with an additional 20 mg dose (that is 40mg total) at both Week 0 and Week 4.
- Placebo: Subject will receive subcutaneous administration of matching placebo of ofatumumab once every 4 weeks through Week 56, with an additional dose at both Week 0 and Week 4.
Period: Overall Study
Arm/Group | Ofatumumab | Placebo
Started | 17 | 18
Requiried Individualized Follow-up | 1 | 0
Completed | 2 | 1
Not Completed | 15 | 17
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Study closed/terminated | 14 | 15
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofatumumab | Placebo | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (8.70) | 47.1 (11.20) | 48.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 7 | 10 | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 0 | 1
  American Indian or Alaskan Native | 1 | 2 | 3
  Asian - East Asian Heritage | 2 | 0 | 2
  Asian - Japanese Heritage | 1 | 1 | 2
  White - Arabic/North African Heritage | 2 | 1 | 3
  White - White/ Caucasian/ European Heritage | 10 | 14 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced Sustained Remission on Minimal Steroid Therapy
Description: Sustained remission = time from randomization to the time of the subject's initial reduction of prednisone/prednisolone dose to <=10 mg/day and maintenance of a dose <=10 mg/day with no new or nonhealing lesions for >=8 weeks and maintenance of the status until Week 60.
Time Frame: Baseline up to approximately 60 weeks
Measure: Number; unit: participants
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 17 | 18
participants | 0 | 0

2. Primary Outcome: Duration of Remission on Minimal Steroid Therapy
Description: Sum of all periods of absence of new or nonhealing lesions while on an oral prednisone/prednisolone dose of <=10 mg/day up to Week 60 was assessed.
Time Frame: Baseline up to approximately 60 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 3 | 1
days | 168.0 (73.33) | 122.0 (NA) — There is only one subject

3. Secondary Outcome: Percentage of Subjects Achieving Remission on Minimal Steroid Therapy at Week 60
Description: Percentage of subjects who achieved absence of new or nonhealing lesions while on an oral prednisone/prednisolone dose of <=10 mg/day for > or = 8 weeks at Week 60 was assessed. Time to remission was not estimable.
Time Frame: Week 60
Measure: Number; unit: percentage of participants
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 17 | 18
percentage of participants | 17.6 | 5.6

4. Secondary Outcome: Time to Remission While on Minimal Steroid Therapy by Week 60.
Description: Time from randomization to the time of the subject's initial reduction of prednisone/prednisolone dose to <=10 mg/day and maintained dose at <=10 mg/day with no new or nonhealing lesions for >=8 weeks by Week 60 was assessed
Time Frame: Baseline up to approximately 60 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 17 | 18
days | NA [57.0 to NA] — Due to limited sample size value is not estimable | NA [NA to NA] — Due to limited sample size value is not estimable

5. Secondary Outcome: Percentage of Subjects Achieving Remission While Off Steroid Therapy by Week 60
Description: Percentage of subjects with initial reduction of all steroids for >=8 weeks with an absence of new or nonhealing (established) lesions by Week 60 were to be assessed. All subjects remained on prednisone/prednisolone so this endpoint could not be analyzed.Time to remission off steroid therapy also could not be analyzed
Time Frame: Baseline up to approximately 60 weeks
Population: All participants remained on steroid therapy
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Days a Subject Maintained Minimal Steroid Therapy by Week 60.
Description: Number of days a subject maintained minimal steroid therapy (an oral prednisone/prednisolone dose of ≤10 mg/day in the absence of new or nonhealing lesions) by Week 60.
Time Frame: Baseline up to approximately 60 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 3 | 1
days | 168 (73.33) | 122.0 (NA) — Only one paraticipant

7. Secondary Outcome: Time to Initial Flare/Relapse by Week 60
Description: Time from randomization to the time of appearance of >=3 new lesions within 1 month that did not heal spontaneously within 1 week, or to the time when there was an extension of lesions that were present at the randomization by Week 60 was assessed
Time Frame: Baseline up to approximately 60 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 2 | 8
days | 448 [NA to NA] — Due to limited sample size values are not estimable | 169.0 [86.0 to 284.0]

8. Secondary Outcome: Percentage of Participants With no Flare/Relapse by Week 60
Description: Percentage of participants achieving absence of new or nonhealing lesions while on an oral prednisone/prednisolone dose of <=10 mg/day and did not subsequently have a appearance of >=3 new lesions within 1 month that did not heal spontaneously within 1 week, or to the time when there was an extension of lesions that were present at the randomization by Week 60 was assessed
Time Frame: Baseline up to approximately 60 weeks
Population: number of participants varied across visits
Measure: Number; unit: percentage of participants
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 17 | 18
percentage of participants
  Week 2 no flare: number analyzed (Participants) | 17 | 17
  Week 2 no flare | 100.0 | 94.4
  Week 2 no new/nonhealing lesions: number analyzed (Participants) | 17 | 17
  Week 2 no new/nonhealing lesions | 47.1 | 22.2
  Week 4 no flare: number analyzed (Participants) | 15 | 16
  Week 4 no flare | 88.2 | 83.3
  Week 4 no new/nonhealing lesions: number analyzed (Participants) | 15 | 16
  Week 4 no new/nonhealing lesions | 47.1 | 38.9
  Week 6 no flare: number analyzed (Participants) | 12 | 15
  Week 6 no flare | 70.6 | 77.8
  Week 6 no new/nonhealing lesions: number analyzed (Participants) | 12 | 15
  Week 6 no new/nonhealing lesions | 41.2 | 33.3
  Week 8 no flare: number analyzed (Participants) | 11 | 14
  Week 8 no flare | 64.7 | 72.2
  Week 8 no new/nonhealing lesions: number analyzed (Participants) | 11 | 14
  Week 8 no new/nonhealing lesions | 35.3 | 33.3
  Week 12 no flare: number analyzed (Participants) | 10 | 12
  Week 12 no flare | 58.8 | 55.6
  Week 12 no new/nonhealing lesions: number analyzed (Participants) | 10 | 12
  Week 12 no new/nonhealing lesions | 35.3 | 16.7
  Week 16 no flare: number analyzed (Participants) | 9 | 12
  Week 16 no flare | 52.9 | 61.1
  Week 16 no new/nonhealing lesions: number analyzed (Participants) | 9 | 12
  Week 16 no new/nonhealing lesions | 23.5 | 16.7
  Week 20 no flare: number analyzed (Participants) | 8 | 12
  Week 20 no flare | 47.1 | 50.0
  Week 20 no new/nonhealing lesions: number analyzed (Participants) | 8 | 12
  Week 20 no new/nonhealing lesions | 29.4 | 16.7
  Week 24 no flare: number analyzed (Participants) | 8 | 11
  Week 24 no flare | 47.1 | 38.9
  Week 24 no new/nonhealing lesions: number analyzed (Participants) | 8 | 11
  Week 24 no new/nonhealing lesions | 35.3 | 16.7
  Week 28 no flare: number analyzed (Participants) | 5 | 7
  Week 28 no flare | 29.4 | 22.2
  Week 28 no new/nonhealing lesions: number analyzed (Participants) | 5 | 7
  Week 28 no new/nonhealing lesions | 17.6 | 11.1
  Week 32 no flare: number analyzed (Participants) | 6 | 6
  Week 32 no flare | 35.3 | 27.8
  Week 32 no new/nonhealing lesions: number analyzed (Participants) | 6 | 6
  Week 32 no new/nonhealing lesions | 17.6 | 5.6
  Week 36 no flare: number analyzed (Participants) | 4 | 3
  Week 36 no flare | 23.5 | 11.1
  Week 36 no new/nonhealing lesions: number analyzed (Participants) | 4 | 3
  Week 36 no new/nonhealing lesions | 5.9 | 5.6
  Week 40 no flare: number analyzed (Participants) | 3 | 2
  Week 40 no flare | 17.6 | 5.6
  Week 40 no new/nonhealing lesions: number analyzed (Participants) | 3 | 2
  Week 40 no new/nonhealing lesions | 11.8 | 0
  Week 44 no flare: number analyzed (Participants) | 3 | 2
  Week 44 no flare | 17.6 | 5.6
  Week 44 no new/nonhealing lesions: number analyzed (Participants) | 3 | 2
  Week 44 no new/nonhealing lesions | 5.9 | 0
  Week 48 no flare: number analyzed (Participants) | 3 | 1
  Week 48 no flare | 17.6 | 0
  Week 48 no new/nonhealing lesions: number analyzed (Participants) | 3 | 1
  Week 48 no new/nonhealing lesions | 0 | 0
  Week 52 no flare: number analyzed (Participants) | 2 | 1
  Week 52 no flare | 11.8 | 5.6
  Week 52 no new/nonhealing lesions: number analyzed (Participants) | 2 | 1
  Week 52 no new/nonhealing lesions | 11.8 | 0
  Week 56 no flare: number analyzed (Participants) | 2 | 1
  Week 56 no flare | 11.8 | 0
  Week 56 no new/nonhealing lesions: number analyzed (Participants) | 2 | 1
  Week 56 no new/nonhealing lesions | 5.9 | 0
  Week 60 no flare: number analyzed (Participants) | 17 | 17
  Week 60 no flare | 88.2 | 83.3
  Week 60 no new/nonhealing lesions: number analyzed (Participants) | 17 | 17
  Week 60 no new/nonhealing lesions | 52.9 | 33.3

9. Secondary Outcome: Plasma Trough Concentrations of Ofatumumab
Description: Only plasma (trough) concentrations of ofatumumab were presented
Time Frame: 4 hours post baseline, Days 1-4,7,14, Weeks 4,8,12,16,20,24,36,48,52,56, up to approximately 60 weeks
Population: number of participants varied across visits
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ofatumumab
Number analyzed (Participants) | 17
ng/mL
  4 hours post dose SS: number analyzed (Participants) | 1
  4 hours post dose SS | 56.60 (NA) — only 1 participant
  Day 1 Steady State (SS): number analyzed (Participants) | 1
  Day 1 Steady State (SS) | 1917.50 (NA) — only 1 participant
  Day 2 Steady State (SS): number analyzed (Participants) | 1
  Day 2 Steady State (SS) | 2994.20 (NA) — only 1 participant
  Day 3 Steady State (SS): number analyzed (Participants) | 1
  Day 3 Steady State (SS) | 3553.80 (NA) — only 1 participant
  Day 4 Steady State (SS): number analyzed (Participants) | 1
  Day 4 Steady State (SS) | 3619.20 (NA) — only 1 participant
  Day 7 Steady State (SS): number analyzed (Participants) | 1
  Day 7 Steady State (SS) | 3434.90 (NA) — only 1 participant
  Day 14 Steady State (SS): number analyzed (Participants) | 1
  Day 14 Steady State (SS) | 2055.30 (NA) — only 1 participant
  Week 4: number analyzed (Participants) | 12
  Week 4 | 311.59 (278.011)
  Week 4 SS: number analyzed (Participants) | 1
  Week 4 SS | 1132.70 (NA) — only 1 participant
  Week 8: number analyzed (Participants) | 9
  Week 8 | 1253.60 (439.574)
  Week 8 SS: number analyzed (Participants) | 2
  Week 8 SS | 1456.95 (668.994)
  Week 12: number analyzed (Participants) | 7
  Week 12 | 727.01 (430.834)
  Week 12 SS: number analyzed (Participants) | 3
  Week 12 SS | 900.00 (455.930)
  Week 16: number analyzed (Participants) | 8
  Week 16 | 512.88 (377.189)
  Week 16 SS: number analyzed (Participants) | 1
  Week 16 SS | 1043.40 (NA) — only 1 participant
  Week 20: number analyzed (Participants) | 6
  Week 20 | 415.88 (303.307)
  Week 20 SS: number analyzed (Participants) | 2
  Week 20 SS | 720.10 (246.356)
  Week 24: number analyzed (Participants) | 5
  Week 24 | 461.72 (437.717)
  Week 24 SS: number analyzed (Participants) | 3
  Week 24 SS | 686.10 (329.699)
  Week 36: number analyzed (Participants) | 3
  Week 36 | 477.63 (378.112)
  Week 36 SS: number analyzed (Participants) | 1
  Week 36 SS | 931.20 (NA) — only 1 participant
  Week 48: number analyzed (Participants) | 2
  Week 48 | 352.95 (300.591)
  Week 48 SS: number analyzed (Participants) | 1
  Week 48 SS | 1230.40 (NA) — only 1 participant
  Week 52 SS: number analyzed (Participants) | 1
  Week 52 SS | 897.30 (NA) — only 1 participant
  Week 56: number analyzed (Participants) | 2
  Week 56 | 436.40 (511.662)
  Week 60: number analyzed (Participants) | 2
  Week 60 | 76.40 (32.244)
  Early withdrawal: number analyzed (Participants) | 12
  Early withdrawal | 925.91 (971.715)

10. Secondary Outcome: Number of Participants With Values Below Lower Limit of Normal for Immunoglobulin A
Description: Assessed by the incidence, titer, and type of human anti-human antibody (HAHA) immune response
Time Frame: Baseline up to approximately 60 weeks
Population: number of participants varied across visits
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 17 | 18
Participants
  Baseline | 1 | 0
  Week 12: number analyzed (Participants) | 10 | 11
  Week 12 | 1 | 0
  Week 16: number analyzed (Participants) | 0 | 1
  Week 16 |  | 0
  Week 24: number analyzed (Participants) | 8 | 11
  Week 24 | 1 | 0
  Week 36: number analyzed (Participants) | 4 | 3
  Week 36 | 1 | 0
  Week 48: number analyzed (Participants) | 3 | 1
  Week 48 | 1 | 0
  Week 52: number analyzed (Participants) | 2 | 1
  Week 52 | 1 | 0
  Week 56: number analyzed (Participants) | 2 | 1
  Week 56 | 1 | 0
  Week 60/Early withdrawal | 0 | 0
  First 12 weeks of therapy | 1 | 0
  During on therapy period | 1 | 0

11. Secondary Outcome: Number of Participants With Values Below Lower Limit of Normal for Immunoglobulin G
Description: Assessed by the incidence, titer, and type of human anti-human antibody (HAHA) immune response
Time Frame: Baseline up to approximately 60 weeks
Population: number of participants varied across visits
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 17 | 18
Participants
  Baseline | 1 | 2
  Week 12: number analyzed (Participants) | 10 | 11
  Week 12 | 0 | 1
  Week 16: number analyzed (Participants) | 0 | 1
  Week 16 |  | 1
  Week 24: number analyzed (Participants) | 8 | 11
  Week 24 | 0 | 1
  Week 36: number analyzed (Participants) | 4 | 3
  Week 36 | 0 | 0
  Week 48: number analyzed (Participants) | 3 | 1
  Week 48 | 0 | 0
  Week 52: number analyzed (Participants) | 2 | 1
  Week 52 | 0 | 0
  Week 56: number analyzed (Participants) | 2 | 1
  Week 56 | 0 | 0
  Week 60/Early withdrawal | 0 | 2
  First 12 weeks of therapy | 1 | 3
  During on therapy period | 1 | 4

12. Secondary Outcome: Number of Participants With Values Below Lower Limit of Normal for Immunoglobulin M
Description: Assessed by the incidence, titer, and type of human anti-human antibody (HAHA) immune response
Time Frame: Baseline up to approximately 60 weeks
Population: number of participants varied across visits
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 17 | 18
Participants
  Baseline | 1 | 1
  Week 12: number analyzed (Participants) | 10 | 11
  Week 12 | 4 | 1
  Week 16: number analyzed (Participants) | 0 | 1
  Week 16 |  | 0
  Week 24: number analyzed (Participants) | 8 | 11
  Week 24 | 4 | 0
  Week 36: number analyzed (Participants) | 4 | 3
  Week 36 | 4 | 0
  Week 48: number analyzed (Participants) | 3 | 1
  Week 48 | 3 | 0
  Week 52: number analyzed (Participants) | 2 | 1
  Week 52 | 2 | 0
  Week 56: number analyzed (Participants) | 2 | 1
  Week 56 | 2 | 0
  Week 60/Early withdrawal | 6 | 2
  First 12 weeks of therapy | 4 | 1
  During on therapy period | 6 | 2

13. Secondary Outcome: Largest Mean Decrease From Baseline for Immunoglobulin A, G and M
Description: Immunoglobulins A, G and M were assessed by the incidence, titer, and type of human anti-human antibody (HAHA) immune response
Time Frame: Baseline up to approximately 60 weeks
Population: number of participants varied across visits
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 17 | 18
g/L
  Immunoglobulin A: number analyzed (Participants) | 13 | 11
  Immunoglobulin A | -0.185 (0.1181) | -0.472 (0.7116)
  Immunoglobulin G: number analyzed (Participants) | 11 | 13
  Immunoglobulin G | -1.172 (0.9390) | -0.955 (0.6205)
  Immunoglobulin M: number analyzed (Participants) | 17 | 11
  Immunoglobulin M | -0.231 (0.1152) | -0.263 (0.3053)

14. Secondary Outcome: Change From Baseline for CD19+ B Cell Count
Description: CD19+ B cell count will be performed using Flow Cytometry
Time Frame: Baseline up to approximately 60 weeks
Population: number of participants varied across visits
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Ofatumumab | Placebo
Number analyzed (Participants) | 17 | 18
10^9 cells/L
  Week 12: number analyzed (Participants) | 10 | 10
  Week 12 | -0.24940 (0.228704) | 0.03080 (0.072358)
  Week 16: number analyzed (Participants) | 0 | 1
  Week 16 |  | 0.08000 (NA) — Not estimable
  Week 24: number analyzed (Participants) | 7 | 9
  Week 24 | -0.28607 (0.265327) | -0.04022 (0.197867)
  Week 36: number analyzed (Participants) | 4 | 3
  Week 36 | -0.20525 (0.052703) | -0.10033 (0.021385)
  Week 48: number analyzed (Participants) | 3 | 1
  Week 48 | -0.19717 (0.061436) | -0.00200 (NA) — Not estimable
  Week 52: number analyzed (Participants) | 2 | 1
  Week 52 | -0.16300 (0.023335) | 0.09600 (NA) — Not estimable
  Week 56: number analyzed (Participants) | 2 | 1
  Week 56 | -0.16300 (0.023335) | 0.01000 (NA) — Not estimable
  Week 60/Early withdrawal | -0.21403 (0.190282) | 0.00367 (0.190375)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 60 months
Groups:
- Ofatumumab SC: Subject will receive subcutaneous administration of ofatumumab 20 mg once every 4 weeks through Week 56, with an additional 20 mg dose (that is 40mg total) at both Week 0 and Week 4.
Arm/Group | Ofatumumab SC | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/18
Other Adverse Events (participants affected / at risk) | 14/17 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab SC (N=17) | Placebo (N=18)
Hepatic enzyme increased (Investigations) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab SC (N=17) | Placebo (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Conjunctival discolouration (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 3 | 0
Fatigue (General disorders) | 2 | 1
Influenza like illness (General disorders) | 1 | 1
Local reaction (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 3 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
B-lymphocyte count decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Persistent depressive disorder (Psychiatric disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Semen discolouration (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-09-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT01920477/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT01920477/SAP_001.pdf